CLINICAL TRIAL: NCT03126669
Title: Oxygen as a Limiting Factor for Performing Multitasking: Functional Evaluation Under Normobaric and Hyperbaric Oxygenation of Healthy Participants
Brief Title: Oxygen as a Limiting Factor for Performing Multitasking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 213/13
Record Dates: First submitted 2017-04-20; First posted 2017-04-24 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Cognitive Change
Keywords: Hyperbaric oxygen; multitasking performance; cognitive funcitons
MeSH Terms: interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treratment (Active Comparator): 100% oxygen at 2 ATA at the hyperbaric chamber
  Interventions: Device: Hyperbaric oxygen
- Placebo (Placebo Comparator): normal air, in the hyperbaric chamber
  Interventions: Device: Hyperbaric chamber, normal air

INTERVENTIONS:
Device: Hyperbaric oxygen — Breathing 100% oxygen at 2ATA in the hyperbaric chamber
  Arms: Treratment
Device: Hyperbaric chamber, normal air — Hyperbaric chamber with normal air
  Arms: Placebo

SUMMARY:
The aim of the present study was to evaluate whether hyperbaric oxygen (HBO) environment, with increased oxygen supply to the brain, will enable better performance of complex and/or multiple activities.

DETAILED DESCRIPTION:
The Brain uses 20% of the total oxygen supply consumed by the entire body. Even though, less than 10% of the brain is active at every given time, the brain utilizes almost all the oxygen delivered. In order to perform different tasks or more than one task (multi-tasking), the oxygen supply is shifted from one brain region to another, via modulation of blood perfusion.

The aim of the present study was to evaluate whether hyperbaric oxygen (HBO) environment, with increased oxygen supply to the brain, will enable better performance of complex and/or multiple activities.

Methods: a prospective, double blind randomized control, cross over trial including healthy volunteers. Participants were asked to perform a cognitive task, a motor task and a simultaneous cognitive-motor task (multi-tasking). Participants were randomized to perform the tasks at 2 environments: (a) normobaric air (1ATA 21% oxygen) (b) HBO (2ATA 100% oxygen). Two weeks later participants were crossed to the alternative environment. Blinding of the normobaric environment was achieved in the same chamber with masks on while hyperbaric sensation was simulated by increasing pressure in the first minute and gradually decreasing to normobaric environment prior to tasks performance.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers,
* minimum of 12 years of formal education

Exclusion Criteria:

* any inner ear pathologies,
* any lung disease,
* any mental or physical limitation of participat in going into oxygen chamber environment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2017-03-25 (Actual)

PRIMARY OUTCOMES:
Cognitive/Attention Symbol-Digit Modality Test (SDMT) | 45 minutes
  Three different forms of the SDMT were used in each evaluation session. The first was a try-out for the test, ensuring understanding of the task. The second tests the ability to per-form an individual task. The third form was used together with the motor test for examin-ing dual task performance. Standard administration procedures were followed as indicat-ed in the test manual. The score of the test is the number of correct substitutions during 90-second interval.
Motor task: transferring of beans | 45 minutes
  Motor performance was evaluated by the Motor Assessment Scale test (MAS) - transfer-ring units of beans one by one between two tea cups an arm length away.

CONTACTS AND LOCATIONS:
Overall Officials: Shai a Efrati, MD, Principal Investigator — Asaf-Harofhe MC
Locations (1):
- Assaf-Harofeh Medical Center, Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: No